CLINICAL TRIAL: NCT03528473
Title: Adapted Physical Activity (APA), Insulin Resistance, Oxidative Stress and Microcirculatory Haemodynamics in Breast Cancer Patients.
Brief Title: Adapted Physical Activity (APA) in a Breast Cancer Population.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Ettore Marini, Resident in Internal Medicine, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APA-PG1
Record Dates: First submitted 2018-03-22; First posted 2018-05-17 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Breast Neoplasms; Exercise; Exercise Therapy; Insulin Resistance; Oxidative Stress; Microcirculation; Quality of Life; Atherosclerosis
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Insulin Resistance; Atherosclerosis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, double-group assignment, open label study with intermediate crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Patients involved in the 6 months-physical training group.
  Interventions: Other: Exercise
- Control (No Intervention): Patients in control group carry on their usual follow-up programme.

INTERVENTIONS:
Other: Exercise — The exercise intervention consists of 60 minutes sessions, divided into 40 minutes of aerobic exercise and 20 minutes of circuit training for muscular strength and flexibility exercises.
  Aerobic exercise is performed using treadmill, exercise bikes, syncro and arm-ergometers, gradually increasing the exercise intensity, after a 10 minutes period of warming-up, to 60-80 % of Maximum Heart Rate.
  Resistance training consists of resistance exercises for large muscle groups, performed with body weight-exercises and isotonic machines.
  Arms: Exercise

SUMMARY:
The aim of this study is to investigate the effect of a 6-months program of Adapted Physical Activity (APA) on lifestyle, physical activity levels, insulin resistance and adipokines, oxidative stress, microcirculatory haemodynamics and serum levels of specific circulating miRNA in post-menopausal, physically inactive breast cancer patients in oncologic follow-up with or without hormone therapy that had completed adjuvant treatment (radiotherapy and/or chemotherapy) .

Furthermore, the study will determine the impact of APA on functional capabilities, on self-reported physical activity, quality of life and psychic health.

DETAILED DESCRIPTION:
This is a randomized controlled double-group assignment study with intermedial switch-over including post-menopausal, physically inactive breast cancer patients in oncological follow-up with or without hormone therapy, that had completed adjuvant post-surgical treatment (radiotherapy and/or chemotherapy) from at least 3 months and from not more than 3 years.

Patients in hormonal therapy and patient not in hormonal therapy will be assigned in two different groups, each one of 50 patients. In each groups, patients will be randomized divided in a control group (25 pt) and in a 6 months-physical training group (25 pt). After 6-months patient in control group will be switched in the physical training group.

The duration of the study is 2 year. Clinical evaluation of the patients will be made: at the enrollment, after 6, 12, and 24 months.

Physical activity will be adapted according to arm and shoulder morbidity, after fracture risk assessment. Exercise will be concentrated solely on leg muscles (pedalling on a cycle or bed ergometer) in individuals with limitations in the range of motion of the arms (eg, due to breast, axillary, or thoracic surgery). In patients experiencing ataxia, dizziness, or peripheral neuropathy, walking outdoors and mostly cycle-ergometry training will be preferred to other activities that also involve large muscle groups but require additional balance and coordination (eg, treadmill walking, outdoor cycling).

Exercises will be performed at the Unipolar Spinal Unit of "S. Maria della Misericordia" Hospital, Perugia.

The aim of the study is to confirm the positive effect of APA on metabolic stress, body mass composition, functional capacity, serum levels of specific circulating miRNA and quality of life in breast cancer patients in oncological follow-up.

Currently, only few data are available about the relationship between physical activity and microcirculatory hemodynamics that, together with oxidative stress, could be involved in genesis and progression of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients in oncological follow-up
* post-menopausal age
* physically inactivity (light to moderate or vigorous leisure-time physical activity less than 10 minutes a day, US National Health Interview Survey)
* assuming or not hormone therapy
* after 3 months - 3 years from adjuvant post-surgical treatment (radiotherapy and/or chemotherapy)

Exclusion Criteria:

Permanent

* Patients older than 80 years
* Inability to carry on physical activity
* Metastatic neoplasia or unknown stage and/or histology
* Concomitant neoplasia
* Patients on corticosteroid treatment
* Known heart disease (heart failure NYHA II (New York Heart Association II) or superior, angina pectoris or positive exercise stress test, treatment-related cardiotoxicity)
* Currently on a weight loss plan or on moderate physical activity before the start of the project (no more than three sessions a week)
* Severe cachexia (loss of more than of 35% premorbid weight or weight loss more than 10% in the last 6 months).
* Morbidly obesity (BMI >40 kg/m2),
* Immunodepression (absolute neutrophils count < 500/mmc)

Temporary

* Uncontrolled pain or new onset bone pain until further diagnostic study
* Severe anemia (haemoglobin below 8 g/dL) or platelet count lower than <50000/μL
* Fever (temperature above 38ºC) or acute infections
* Severe nausea and vomiting within previous 24-36 h
* Uncontrolled blood pressure (systolic blood pressure > 160 mm Hg and/or diastolic blood pressure >99 mm Hg)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity levels | Evaluation baseline and after 6, 12 and 24 months from enrollment.
  Self reported physical activity, using IPAQ-SF (International Physical Activity Questionnairev - Short Form) score
Change in BMI | Evaluation baseline and after 6, 12 and 24 months from enrollment.
  Reduction of BMI expressed as body mass (kg) / height^2 (m^2)

SECONDARY OUTCOMES:
Change in Post-Occlusive Reactive Hyperemia (PORH) | Evaluation baseline and after 6, 12 and 24 months from enrollment.
  Improvement of Area of Hyperemia (AH) at Post-Occlusive Reactive Hyperemia (PORH) on Laser Doppler velocimetry (Periflux System 5000, Perimed), expressed as Perfusion Units (PU).
Carotid intima-media thickness (IMT) | Evaluation baseline and after 6, 12 and 24 months from enrollment.
  Improvement of macrovascular structures, that will be explored by carotid intima-media thickness (IMT) (two-dimensional B-mode ultrasonography), measured in mm.
Arterial stiffness | Evaluation baseline and after 6, 12 and 24 months from enrollment.
  Reduction of arterial stiffness, that will be evaluated by radial applanation tonometry (SphygmoCor) and general transfer function assessing PWV (measure in m/s).
Hemorheological profile | Evaluation baseline and after 6, 12 and 24 months from enrollment.
  Improvement of Hemorheological profile, that will be studied with Serum, Plasma, and Blood Viscosity (Haake rotational viscometer), measured as mPas.
Serum adiponectin | Evaluation baseline and after 6, 12 and 24 months from enrollment.
  Improvement of serum adiponectin, measured by ELISA-method (ng/ml). Blood samples will be collected in the morning between 7:00 and 9:00 am, after overnight fasting.
Serum IGF-1 | Evaluation baseline and after 6, 12 and 24 months from enrollment.
  Improvement of serum IGF-1, measured by ELISA-method (ng/ml). Blood samples will be collected in the morning between 7:00 and 9:00 am, after overnight fasting.
VFA (Visceral Fat Area) | Evaluation baseline and after 6, 12 and 24 months from enrollment.
  Improvement of Ultrasound assesment of visceral fat area (VFA, by MyLab 50 Ultrasonography, Esaote), measured by Hirooka formula (cm^2)
HOMA-IR index | Evaluation baseline and after 6, 12 and 24 months from enrollment.
  Homeostatic model assessment (HOMA) for insulin resistance (IR) is a method for assessing β-cell function and insuline resistance from basal (fasting) glucose and insulin or C-peptide concentrations. HOMA-IR can be calculated with a simple mathematical approximation as HOMA-IR = (FPI × FPG)/22.5, where FPI is fasting plasma insulin concentration (mU/l) and FPG is fasting plasma glucose (mmol/l), or as HOMA-IR = (FPI × FPG)/405 if fasting plasma glucose is expressed in mg/dl.
  Values bethween 3 and 5 are considered expression of moderate insuline resistance; values upper 5 are considered expression of severe insuline resistance.
  Improvement of insulin-sensitivity expressed as HOMA-IR index reduction.
Maximal aerobic capacity (VO2max) | Evaluation baseline and after 6, 12 and 24 months from enrollment.
  Increase of maximal aerobic capacity after physical training, measured as ml/kg/min.
miRNA | Evaluation baseline and after 6, 12 and 24 months from enrollment.
  Variation of serum miR-10b, 15a, 146, 155, 375 e let-7a,b,c concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Leonella Pasqualini, MD, Study Director — University Of Perugia
Locations (1):
- University of Perugia, Perugia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adraskela K, Veisaki E, Koutsilieris M, Philippou A. Physical Exercise Positively Influences Breast Cancer Evolution. Clin Breast Cancer. 2017 Oct;17(6):408-417. doi: 10.1016/j.clbc.2017.05.003. Epub 2017 May 19. PMID 28606800
- [Background] Foucaut AM, Berthouze-Aranda SE, Touillaud M, Kempf-Lepine AS, Baudinet C, Meyrand R, Carretier J, Bachmann P, Fervers B. Reduction of health risk factors through an adapted physical activity program in patients with breast cancer. Support Care Cancer. 2014 Apr;22(4):1097-104. doi: 10.1007/s00520-013-2065-3. Epub 2013 Dec 3. PMID 24292096
- [Background] Franses JW, Edelman ER. The evolution of endothelial regulatory paradigms in cancer biology and vascular repair. Cancer Res. 2011 Dec 15;71(24):7339-44. doi: 10.1158/0008-5472.CAN-11-1718. Epub 2011 Dec 5. PMID 22144472
- [Background] Ye J, Jia J, Dong S, Zhang C, Yu S, Li L, Mao C, Wang D, Chen J, Yuan G. Circulating adiponectin levels and the risk of breast cancer: a meta-analysis. Eur J Cancer Prev. 2014 May;23(3):158-65. doi: 10.1097/CEJ.0b013e328364f293. PMID 23929213
- [Background] Tesarova P, Kalousova M, Zima T, Suchanek M, Malikova I, Kvasnicka J, Duskova D, Tesar V, Vachek J, Krupickova-Kasalova Z, Malik J. Endotelial activation and flow-mediated vasodilation in young patients with breast cancer. Neoplasma. 2013;60(6):690-7. doi: 10.4149/neo_2013_088. PMID 23906304